CLINICAL TRIAL: NCT03534726
Title: Edema and Fibrosis Cardiac Magnetic Resonance Imaging in Cardiomyopathy
Brief Title: Edema and Fibrosis CMR Imaging in Cardiomyopathy
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 827516
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Patients: Patients with cardiomyopathy
  Interventions: Device: 7 T CMR
- Normal subjects: No prior history of heart disease.
  Interventions: Device: 7 T CMR

INTERVENTIONS:
Device: 7 T CMR — 7 tesla MRI device

SUMMARY:
7 Tesla MRI is a new magnetic field strength that has become available at Penn for cardiovascular MRI. This new scanner has potential to improve assessment of cardiovascular disease due to its increased signal-to-noise ratio, higher spatial resolution, and response to magnetic properties of tissue at high field. The purpose of this study is to assess the feasibility of 7 T CMR. Secondly, we wish to investigate its use, to improve clinical and research MRI. Altogether, 7 T may permit better clinical diagnosis of cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 20-70 years old

Exclusion Criteria:

* Advanced renal disease (estimated GFR rate < 30 mL/min) or hypersensitivity to gadolinium contrast agent.
* Presence of cardiac pacemaker or implanted cardioverter defibrillator
* Pregnancy
* Inability to provide informed consent
* Other contraindications to MRI (such as claustrophobia)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The eligible population are cardiomyopathy patients and normal volunteers.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ejection fraction | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided